CLINICAL TRIAL: NCT02556320
Title: Immunological and Viral Parameters in Patients Receiving Anti-epileptic Drugs
Acronym: VIRIDAE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012/075/HP
Record Dates: First submitted 2015-09-18; First posted 2015-09-22 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Epilepsy; Drug Hypersensitivity Syndrome
MeSH Terms: conditions — Epilepsy; Drug Hypersensitivity Syndrome | interventions — Anticonvulsants; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Epileptic patient (Experimental): Blood sampling is done for Patient who initiate anti-epileptic drug (sodium valproate, divalproate sodium, valpromide, lamotrigine, carbamazepine, oxcarbazepine, eslicarbazepine acetate)
  Interventions: Drug: anti-epileptic drug; Biological: Blood sampling

INTERVENTIONS:
Drug: anti-epileptic drug — Patient who initiate anti-epileptic drug (sodium valproate, divalproate sodium, valpromide, lamotrigine, carbamazepine, oxcarbazepine, eslicarbazepine acetate)
Biological: Blood sampling — Blood sampling is done for Patient who initiate anti-epileptic drug (sodium valproate, divalproate sodium, valpromide, lamotrigine, carbamazepine, oxcarbazepine, eslicarbazepine acetate)

SUMMARY:
A recent study has shown that certain drug allergies were actually related to an immune system against certain viruses. The aim of the study is to evaluate, in patients taking antiepileptic drugs, if this treatment induces proliferation of these viruses and secondarily an immune response that would promote the development of a rash. In particular, will be studied whether these drugs can induce virus reactivation "dormant" in the immune system. This study will not affect the usual follow-up proposed by investigators, with the exception of some additional blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Patients age over 18 years
* Patient for whom treatment of antiepileptic class will be started or was set for less than 48 hours and including one of the following molecules (as princeps or generic equivalent form): sodium valproate, divalproate sodium, valpromide, lamotrigine, carbamazepine, oxcarbazepine eslicarbazepine acetate.
* Patient or patient's representative who was informed and signed the consent form
* Effective contraception in women of childbearing age
* Affiliation to health insurance

Exclusion Criteria:

* Immunosuppressive therapy in progress or acquired immunodeficiency
* Patient with meningitis or meningoencephalitis
* Patient with known contraindications to any molecules indicated in the study
* Major Patient protection (guardianship) or deprived of liberty by judicial or administrative decision.
* Patient participating in another clinical trial or participated in another trial in the month before.
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-05; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with viral reactivation of Epstein-Barr Virus | 3 Months
  Number of patients with viral reactivation of Epstein-Barr Virus is evaluated in patients initiating an anti-epileptic treatment
Number of patients with viral reactivation of Human Herpes Virus 6 | 3 Months
  Number of patients with viral reactivation of Human Herpes Virus 6 is evaluated in patients initiating an anti-epileptic treatment
Number of patients with viral reactivation of Human Herpes Virus 7 | 3 Months
  Number of patients with viral reactivation of Human Herpes Virus 7 is evaluated in patients initiating an anti-epileptic treatment

SECONDARY OUTCOMES:
Change from baseline in lymphocyte population count | 3 Months
  Lymphocyte population count will be compared between baseline and 3 months after the treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Sophie DUVERT-LEHEMBRE, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France